CLINICAL TRIAL: NCT03695081
Title: Patient Pathway Pharmacist: Drug Optimisation for Hip Fracture Patients - Facilitating a Safe Patient Handover: a Descriptive Study
Brief Title: Patient Pathway Pharmacist - Optimal Drug-related Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Hospital Pharmacy Enterprise, South Eastern Norway (Other)
Responsible Party: Principal Investigator, Ben Tore Henriksen, Clinical Pharmacist, Sykehuset i Vestfold HF
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 59475
Record Dates: First submitted 2018-09-11; First posted 2018-10-03 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hip Fractures; Aging; Patient Fall
Keywords: Medicine review; Patient handoff; Patient hand over; Intertrochanteric fractures; Trochanteric fractures; Subtrochanteric fractures; Hospital readmission; Hospital readmissions; Injuries, Hip; Hospitalization; Hospitalisation; Hip; Fracture; Femoral fractures; Femoral neck fractures; Medication errors; Medication review; Medication reconciliation
MeSH Terms: conditions — Hip Fractures; Hip Injuries; Fractures, Bone; Femoral Fractures; Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: An intervention group is compared to a cross-sectional retrospective group.
  A group of 60 patients with hip fracture will get an intervention by a clinical pharmacist who performs medication reconciliation and medication review during hospitalisation, they will receive a discharge summary where the medication part is optimised. After six weeks the patients will be get a follow-up with a second medication reconciliation and - review. This group will be compared with the last 50 patients with hip fracture who did not get the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Pathway Pharmacist intervention (Experimental): 1. Medication reconciliation at admission to hospital
  2. Medication review post surgery
  3. Optimised list of drugs in the discharge summary, in accordance with hospital procedures
  4. Medication reconciliation, six weeks after discharge
  5. Medication review, six weeks after discharge
  Interventions: Procedure: Patient Pathway Pharmacist intervention
- No intervention (No Intervention): Business as usual. The Patient Pathway Pharmacist is not involved and the nurses and physicians are responsible for medicine reconciliation, -review and section in the discharge summary.

INTERVENTIONS:
Procedure: Patient Pathway Pharmacist intervention — 1. Medication reconciliation at admission to hospital
  2. Medication review post surgery
  3. Optimised list of drugs in the discharge summary, in accordance with hospital procedures
  4. Medication reconciliation, six weeks after discharge
  5. Medication review, six weeks after discharge
  Arms: Patient Pathway Pharmacist intervention

SUMMARY:
Medication errors represent the most common cause of patient injury and one of the most frequently reported health related deviation in Norway. The addition of a dedicated clinical pharmacist throughout the hip fracture patient pathway (patient pathway pharmacist) is believed to improve patient safety and ensure optimal drug-related patient care. The pharmacist will perform medication reconciliation at admission to hospital, medication review after surgery and assist physicians with discharge summary. Six weeks after discharge the patient pathway pharmacist will perform a second drug reconciliation and medication review. This study will assess the pharmacists' place and specific tasks in the patient pathway, describe areas where the pharmacist contribute to increased quality of care and assess the benefits and/or disadvantages experienced with introducing a patient pathway pharmacist. The estimated number of patients included is 60. Current practice will be determined by investigating the last 50 patients' medical record and a questionnaire to health care professionals involved in treatment of hip fracture patients. Data from medication reconciliation and drug review will be collected and compared to current practice. After the inclusion period, focus group surveys and/or semi-structured interviews will be executed to describe the perceived improvement in the quality of care. Primary endpoints are: 1) Medication reconciliation score at admission 2) Number of inappropriate drugs for elderly 3) Discharge summary score 4) Discharge summaries following procedure. Secondary endpoints are readmissions and mortality after 30 and 90 days. Qualitative endpoints: 1) Health care professionals experience of current drug-related practice 2) Experienced advantages and disadvantages of a patient pathway pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture patients in Vestfold county, Norway

Exclusion Criteria:

* Patients under 18 years
* Terminally ill
* Hip fracture patients who do not follow the standardized patient pathway at Vestfold Regional Hospital
* Patients who do not consent to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Discharge summary score | At discharge (estimated five days after fracture/inclusion)
  In the discharge summary, the section describing drugs is scored in accordance with the national patient safety program
Admission summary score | At hospital admission (estimated to be within 24 hours after fracture)
  In the admission summary, the section describing drugs is scored. The score is adjusted from the discharge summary score to fit the admission note.
Discharge summaries written in accordance with procedure | At discharge (estimated five days after fracture/inclusion)
  In the discharge summary, the section describing drugs should be in accordance with procedure.
Number of inappropriate drugs at discharge | During hospitalisation, after surgery (estimated to be within five days after fracture/inclusion)
  After surgery the medication review may reduce the number of inappropriate drugs (on the STOPP-list).

SECONDARY OUTCOMES:
Readmission | 30 days after discharge
  Patients who are readmitted to hospital is quantified
Readmission | 90 days after discharge
  Patients who are readmitted to hospital is quantified
Death | 30 days after discharge
  The number patients who dies is quantified
Death | 90 days after discharge
  The number of patients who dies is quantified

OTHER OUTCOMES:
Experience of current practice | Prior to or during the early start of the intervention
  A questionnaire will be distributed to all health care professionals involved in the treatment of hip fracture patients
Experience of patient pathway pharmacist | Within three months after last included patient
  Focus groups or semi-structured interviews will be performed to assess the advantages and/or disadvantages of introducing a patient pathway pharmacist.

CONTACTS AND LOCATIONS:
Locations (1):
- Vestfold Hospital Trust, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henriksen BT, Krogseth M, Andersen RD, Davies MN, Nguyen CT, Mathiesen L, Andersson Y. Clinical pharmacist intervention to improve medication safety for hip fracture patients through secondary and primary care settings: a nonrandomised controlled trial. J Orthop Surg Res. 2023 Jun 13;18(1):434. doi: 10.1186/s13018-023-03906-2. PMID 37312222
- See also: Score of the drug section in discharge summaries - The Norwegian Patient Safety Programme: In Safe Hands — https://www.itryggehender24-7.no/reduser-pasientskader/legemiddelrelaterte-skader/legemiddelsamstemming-og-legemiddelgjennomgang/_/attachment/download/33b5eb0c-4f62-4d42-862f-b9f95f09423c:12bcc5de3b8e1ff2e4bdb9937951300d8d6f35cc/tiltakspakke-for-samstemming-av-legemiddellister.pdf